CLINICAL TRIAL: NCT01397305
Title: An Extended Feasibility Phase I/II Study of Methylenetetrahydrofolate and Pemetrexed Single Agent, Given as Neoadjuvant Treatment in Patients With Resectable Rectal Cancer
Brief Title: An Extended Feasibility Phase I/II Study of Methylenetetrahydrofolate (Arfolitixorin) and Pemetrexed Single Agent, Given as Neoadjuvant Treatment in Patients With Resectable Rectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Isofol Medical AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISO-MC-091
Record Dates: First submitted 2011-05-25; First posted 2011-07-19 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Rectal Cancer
Keywords: 5,10-methylenetetrahydrofolate; neoadjuvant therapy; pemetrexed; Neoplasms; Rectal Neoplasms; Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Rectal Diseases; Digestive System Diseases; Gastrointestinal Diseases; Intestinal Diseases; Pharmacologic Actions; Therapeutic Uses; Antineoplastic Agents; Enzyme Inhibitors; Molecular Mechanisms of Pharmacological Action; Folic Acid Antagonists; Antimetabolites, Antineoplastic; Antimetabolites
MeSH Terms: conditions — Rectal Neoplasms; Neoplasms; Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Rectal Diseases; Digestive System Diseases; Gastrointestinal Diseases; Intestinal Diseases | interventions — 5,10-methylenetetrahydrofolic acid; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Modufolin and Pemetrexed (Experimental): Modufolin ( [6R] 5,10-methylenetetrahydrofolate) and Pemetrexed
  Interventions: Drug: [6R] 5,10-methylenetetrahydrofolate (arfolitixorin); Drug: Pemetrexed

INTERVENTIONS:
Drug: [6R] 5,10-methylenetetrahydrofolate (arfolitixorin) — 10, 50, 100, 200, and 500 mg/m2 IV on day 1, day 8 day and day 15 of each 21-day cycle. 3 cycles.
  Other Names: Modufolin; 6R-MTHF; ISO-901; arfolitixorin
Drug: Pemetrexed — 500 mg/m2 IV on day 1 of each 21-day cycle. 3 cycles.
  Other Names: ly 231514; multitargeted antifolate

SUMMARY:
The purpose of this study is to determine whether an optimal dose of [6R] 5,10-methylenetetrahydrofolate (arfolitixorin) in combination with pemetrexed are effective in pre-operative treatment of patients with resectable rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathological/ cytological diagnosis of adenocarcinoma of the rectum. Patients must have operable rectal cancer that is amenable to surgery.
* No prior therapy for rectal cancer
* Eastern Cooperative Oncology Group (ECOG) Performance status 0 or 1
* Adequate organ function
* Patient compliance and geographic proximity that allow adequate follow-up
* For women: Must be surgically sterile, postmenopausal, or compliant with a medically approved contraceptive regimen during and for 3 months after treatment; must have a negative serum or urine pregnancy test and must not be lactating.
* For men: Must be surgically sterile or compliant with a contraceptive regimen during and for 3 months after treatment.
* Estimated life expectancy of at least 12 weeks
* Signed informed consent
* At least 18 years of age

Exclusion Criteria:

* Concurrent administration of any other anti-tumor therapy.
* Treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Serious concomitant systemic disorders (e.g., active infection including HIV, cardiac disease) that in the opinion of the investigator would compromise the patient's ability to complete the study.
* Have previously completed or withdrawn from this study or any other study investigating pemetrexed.
* Are pregnant or breast-feeding.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* History of significant neurological or mental disorder, including seizures or dementia.
* Inability to interrupt aspirin or other nonsteroidal anto-inflammatory drugs (NSAIDs)
* Presence of clinically relevant third-space fluid collection that cannot be controlled by drainage or other procedures prior to study entry.
* Inability or unwillingness to be given 5,10-methylenetetrahydrofolate, vitamin B12 or dexamethasone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-04-14 (Actual); Primary Completion 2014-10-16 (Actual); Study Completion 2014-10-16 (Actual)

PRIMARY OUTCOMES:
Feasibility of Pemetrexed Prior to Surgery | 3 cycles (21-day cycles)
  Feasibility is defined as the ability to receive the total planned dose of pemetrexed (i.e., 1500 mg/m) administered over a period of no more than 9 weeks. Feasibility is measured as absence of the following toxicities:
  1. CTC grade 4 lasting >= 7 days, or febrile neutropenia
  2. CTC grade 4 thrombocytopenia or grade 3 with bleeding.
  3. CTC grade 3 nonhematologic toxicity (excluding nausea and vomiting, isolated CTC grade 3 ALT or AST that returns to the patient's pretreatment CTC grade within 3 weeks, or grade 3 fatigue lasting <7 days).

SECONDARY OUTCOMES:
Pathological Complete Response (pCR) | Surgery following 3 cycles (21-day cycles) of chemotherapy
Number of Participants Receiving Sphincter Saving Surgery | Surgery following 3 cycles (21-day cycles) of chemotherapy
Evaluation of qualitative and quantitative toxicities | Start of study treatment until last postoperative visit. Expected average 16 weeks.
  Bleeding, anastomosis, leakage, serious infection.
[6R] 5,10-methylenetetrahydrofolate tissue concentration determination | Surgery following 3 cycles (21-day cycles) of chemotherapy
Correlation between 5,10-methylenetetrahydrofolate and HCy levels in blood | Samples taken prior before study treatment, during 3 cycles of chemotherapy and after completion of study treatment. Expected average 20 weeks.
  Blood samples are taken before start of study treatment, in conjunction with start of every study drug cycle, and after completed study treatment. HCy measurements performed using HPLC. 5-10-methylenetetrahydrofolate is measured in tissue biopsies (tumor and adjacent mucosa) sampled in conjunction with surgery. The tissue is collected before start of study treatment, during and after completed study treatment. 5,10-methylenetetrahydrofolate levels are measured using LC/MS/MS.
Correlation of folate gene polymorphisms and gene signature profiling with clinical outcome and toxicity profiles. | Tissue to be collected from tumor and adjacent mucosa before start of study treatment, during and after completed study treatment. Expected average 20 weeks.
  RT-PCR will be used to measure and determine the gene expression levels of the genes FPGS (Folylpolyglutamate synthase) and GGH (Gamma-glutamyl hydrolase). This translational research will be compared with the clinical outcome and toxicity profiles of patients.
Pharmacokinetic parameters of [6R] 5,10-mTHF, 5-formyl-THF, 5-methyl-THF and THF calculated from plasma | Calculated on Day1 and Day15 after cycle 1 and 3
  Plasma samples will be collected prior to study treatment, and at 10 minutes, 1, 2 and 4 hours after study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bengt G Gustavsson, PhD, MD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden